CLINICAL TRIAL: NCT00184509
Title: Continued Early Intervention for Recent-onset Schizophrenia. A Randomized Controlled Study.
Brief Title: Continued Early Intervention for Recent-onset Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHDIR-1992-1995; NFR-1997-1999
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; psychosocial treatment; outcome
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Behavioral: integrated psychosocial treatment (behavior)

SUMMARY:
The purpose of this study was to determine whether outreach integrated treatment of first episode schizophrenia was more effecive than standard outpatient treatment.

DETAILED DESCRIPTION:
Early intervention for schizophrenia has spawned considerable enthusiasm among clinicians without solid research evidence to suport its benefits and costs. The present study is a random-controlled study of integrated biomedical and psychosocial treatment on a population of recent-onset cases.

Comparison(s): 50 consecutive referrals with schizophrenic disorders of less than two years duration were allocated randomly to a comprehensive model of integrated treatment or standard care for two years. Main outcome measures was psychopathology, psychosocial functioning and hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* first-episode schizophrenia

Exclusion Criteria:

* acute psychosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 1993-02; Study Completion 1998-05

PRIMARY OUTCOMES:
Rehospitalizations and psychotic relapse at two years

SECONDARY OUTCOMES:
Psychopathology, psychosocial changes, functioning, antipsychotic medication

CONTACTS AND LOCATIONS:
Overall Officials: K. Gunnar Gøtestam, MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Derived] Sigrunarson V, Grawe RW, Lydersen S, Morken G. Predictors of long term use of psychiatric services of patients with recent-onset schizophrenia: 12 years follow-up. BMC Psychiatry. 2017 Jan 14;17(1):18. doi: 10.1186/s12888-016-1186-x. PMID 28088223
- [Derived] Sigrunarson V, Grawe RW, Morken G. Integrated treatment vs. treatment-as-usual for recent onset schizophrenia; 12 year follow-up on a randomized controlled trial. BMC Psychiatry. 2013 Jul 30;13:200. doi: 10.1186/1471-244X-13-200. PMID 23898805
- [Derived] Morken G, Widen JH, Grawe RW. Non-adherence to antipsychotic medication, relapse and rehospitalisation in recent-onset schizophrenia. BMC Psychiatry. 2008 Apr 30;8:32. doi: 10.1186/1471-244X-8-32. PMID 18447935
- [Derived] Morken G, Grawe RW, Widen JH. Effects of integrated treatment on antipsychotic medication adherence in a randomized trial in recent-onset schizophrenia. J Clin Psychiatry. 2007 Apr;68(4):566-71. doi: 10.4088/jcp.v68n0409. PMID 17474812